

# Effect of probenecid on synovial fluid ATP levels in CPPD

PROTOCOL AND STATISTICAL ANALYSIS PLAN: NCT02243631

FEBRUARY 28, 2022

# Study protocol

- 1. Subjects diagnosed with CPDD according to the McCarty-Ryan criteria are identified through the rheumatolgy clinical practice.
- 2. Inclusion/Exclusion criteria are met.
- 3. Subjects are interested in participating in the study and sign an informed consent form and HIPPA.
- 4. The affected joint is aspirated for 1 cc of synovial fluid, which is immediately placed on ice and sent to the laboratory for analysis of ATP levels
- 5. The subject is randomized to receive no additional treatment or to receive 2 grams/day of probenecid given in two divided doses.
- 6. The subject is called daily to monitor symptoms in the affected joint and any side effects.
- 7. The subject is seen again by the study team on day 6. Another 1 ml sample of synovial fluid is removed from the affected joint and sent to the laboratory for ATP analysis. The subject is then offered an intra-articular corticosteroid injection in the affected joint.
- 8. This completes the study.

# ATP measurement in Synovial Fluid

### Basal Salt Solution pH 7.5

130 mM NaCl 5 mM KCl 1.5 mM CaCl<sub>2</sub> 1 mM MgCl<sub>2</sub> 5 mM Glucose 0.1% BSA

Mix and then check pH, adjust with NaOH

ATP substrate (FL-AAM from Sigma): Add 5 mL water to vial according to manufacturer's directions.

For standard curve: dilute ATP substrate in salt solution in a ratio of 40% substrate and 60% salt solution. Add 25  $\mu$ l/well for the standard curve.

Standard curve uses the following concentrations of ATP. (1 nM, 2.5 nM, 5 nM, 10 nM, 25 nM, 50 nM, 100 nM)

100  $\mu$ l of salt solution is added to the first well to serve as the zero. 100  $\mu$ l of each of the concentrations of ATP

To Measure the synovial fluid (SF): 100  $\mu$ l of SF (fresh or in citrate) is added to each of 3 wells and then 4  $\mu$ l of the stock ATP substrate is added to the wells. Tap the plate on the counter to mix then read immediately in a plate reader set for luminescence.

N.B. Synovial fluid needs to be measured within 1 hour of collection to avoid loss of ATP.

### **Statistical Analysis Plan**

The primary outcome will be ATP levels measured from extracted synovial fluid. The two treatment groups include those who received probenecid and those with no intervention. A baseline measurement will be taken at the beginning of the study period and another measurement taken at 7 days. Each participant will serve as their own control. A delta will be calculated (7-day ATP level – baseline ATP level) for each participant and a non-parametric Mann-Whitney t-test will be performed. ATP levels commonly require non-parametric analysis as it tends not to be normally distributed. The mean change between baseline and the 7-day timepoint along with the corresponding 95% confidence interval will be presented.

A Wilcoxon matched pairs t-test will be used to assess whether the intervention produced a statistical difference between the two timepoints with probenecid treatment.